CLINICAL TRIAL: NCT03265600
Title: MINDFUL-PC: Integrating Mindfulness Into the Patient-Centered Medical Home - A Comparative Effectiveness Trial of Chronic Illness Self-Management and Action Plan Initiation Among Primary Care Patients
Brief Title: Integrating Mindfulness Into the Patient-Centered Medical Home (Phase 2)
Acronym: MINDFUL-PC-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge Health Alliance (Other)
Collaborators: The Arthur Vining Davis Foundations (Unknown); The Arnold P. Gold Foundation (Other); National Institutes of Health (NIH) (NIH); Brown University (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHA-IRB-1002/08/14_2; UH2AT009145 (NIH)
Record Dates: First submitted 2017-08-28; First posted 2017-08-29 (Actual); Results first posted 2019-12-03 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Depression; Anxiety; Stress Related Disorder; Adjustment Disorders
MeSH Terms: conditions — Depression; Anxiety Disorders; Adjustment Disorders | interventions — Primary Health Care

STUDY DESIGN:
Intervention Model Description: Two arms, intervention and low-dose comparator, which are randomly assigned at the same time and are implemented in parallel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Training for Primary Care (Active Comparator): Mindfulness Training for Primary Care (MTPC) is a primary care adaptation that includes core common Mindfulness-Based Intervention (MBI) elements integrated with novel mindfulness-oriented behavior change elements into a format that is adaptable to delivery in primary care health centers.
  Interventions: Behavioral: Mindfulness Training for Primary Care
- Low-dose Comparator (Other): Comparator arm: Participants receive a 60-minute introduction to mindfulness group plus referral to a list of community mindfulness resources such as private-pay community mindfulness classes, mobile mindfulness applications, books, and online recordings. These participants are added to a 6-month wait-list for a Cambridge Health Alliance mindfulness-based intervention group and allowed to receive behavioral and medical referrals and treatment as usual. All participants complete an action planning protocol during Week 7.
  Interventions: Behavioral: 60-minute Introduction to Mindfulness

INTERVENTIONS:
Behavioral: Mindfulness Training for Primary Care — MTPC is a referral-based, insurance-reimbursable 8-week program that can be delivered as group psychotherapy by Patient-Centered Medical Home-integrated behavioral clinicians or as an 8-week primary care group visit delivered by a primary care provider. MTPC groups are 2 hours long for 8 weeks with a 7-hour weekend day of silent practice. MTPC emphasizes mindfulness-oriented skills for self-regulation, self-management of chronic illness, and health behavior change. All participants complete an action planning protocol during Week 7.
  Arms: Mindfulness Training for Primary Care
Behavioral: 60-minute Introduction to Mindfulness — Participants in the low-dose comparator arm receive a 60-minute introduction to mindfulness. Participants are introduced to the definition(s) of mindfulness, brief mindfulness practices, discussion, and an orientation to an 8-week mindfulness group. They are also given a list of leading community, online, print, and smartphone mindfulness resources.
  Arms: Low-dose Comparator

SUMMARY:
Among primary care patients, compare the effectiveness of an 8-week mindfulness-based intervention (Mindfulness Training for Primary Care[MTPC]) vs. a low-dose mindfulness introduction comparator on self-management of chronic illness and illness-related health behavior action plan initiation, as well as on measures related to anxiety, depression, and stress.

DETAILED DESCRIPTION:
This study builds on a pilot study that investigated the impact of Mindfulness Training for Primary Care on anxiety, depression, stress, and chronic illness self-management in primary care patients receiving care in an urban, community, multi-cultural safety net healthcare system. The current comparative effectiveness randomized controlled trial takes place in a larger sample, and investigates the impact of a refined MTPC curriculum on specific aspects of self-regulation such as action plan initiation, while examining potential mechanisms of change, including self-efficacy, perceived control, mindfulness, self-compassion, emotion regulation, and body awareness. Participants randomized to MTPC are compared with participants who are randomized to a low-dose comparator condition and receive a 1-hour introduction to mindfulness with a referral to community mindfulness resources. Outcome assessments are conducted at baseline and study weeks 8-10.

ELIGIBILITY:
Inclusion Criteria:

* Current CHA patient with an enrolled CHA primary care doctor.
* CHA patients 18 years of age and older.
* Able to tolerate and participate in interviews and engage in all procedures.
* Able to give written consent in English OR willing and able to provide consent and complete assessments through a professional language translator when necessary.
* Diagnosis eligible to be covered by insurance for group visits (e.g., anxiety disorder, depression, or adjustment disorder related to chronic illness, pain, etc.).

Exclusion Criteria:

* Any cognitive impairment that precludes informed consent.
* Patients who, in the opinion of the Principal Investigator, pose an imminent risk of suicide or danger to self or others.
* Likelihood of potential incarceration such as a conviction or pending charges that may potentially result in imprisonment.
* Previous enrollment or randomization of treatment in the present study within the 12 months.
* Behaviors that may cause disruption to a mindfulness group.
* Patients with symptoms of psychosis, thought disorder, and/or severe mental illness, including schizophrenia, schizoaffective, bipolar disorder, or a current severe episode of major depressive disorder.
* Lack of insurance coverage for group psychotherapy may preclude participation in groups.
* Patients in their third trimester of pregnancy who foresee conflicts that preclude their commitment to completing all activities.
* Patients with highly unstable medical problems that put them at a high risk of hospitalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2020-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zev D Schuman-Olivier, MD, Principal Investigator — Cambridge Health Alliance
Locations (1):
- Cambridge Health Alliance, Somerville, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Demarzo MM, Montero-Marin J, Cuijpers P, Zabaleta-del-Olmo E, Mahtani KR, Vellinga A, Vicens C, Lopez-del-Hoyo Y, Garcia-Campayo J. The Efficacy of Mindfulness-Based Interventions in Primary Care: A Meta-Analytic Review. Ann Fam Med. 2015 Nov;13(6):573-82. doi: 10.1370/afm.1863. PMID 26553897
- [Background] Mccubbin T, Dimidjian S, Kempe K, Glassey MS, Ross C, Beck A. Mindfulness-based stress reduction in an integrated care delivery system: one-year impacts on patient-centered outcomes and health care utilization. Perm J. 2014 Fall;18(4):4-9. doi: 10.7812/TPP/14-014. PMID 25662520
- [Background] Sundquist J, Lilja A, Palmer K, Memon AA, Wang X, Johansson LM, Sundquist K. Mindfulness group therapy in primary care patients with depression, anxiety and stress and adjustment disorders: randomised controlled trial. Br J Psychiatry. 2015 Feb;206(2):128-35. doi: 10.1192/bjp.bp.114.150243. Epub 2014 Nov 27. PMID 25431430
- [Background] Merkes M. Mindfulness-based stress reduction for people with chronic diseases. Aust J Prim Health. 2010;16(3):200-10. doi: 10.1071/PY09063. PMID 20815988
- [Background] Goyal M, Singh S, Sibinga EM, Gould NF, Rowland-Seymour A, Sharma R, Berger Z, Sleicher D, Maron DD, Shihab HM, Ranasinghe PD, Linn S, Saha S, Bass EB, Haythornthwaite JA. Meditation programs for psychological stress and well-being: a systematic review and meta-analysis. JAMA Intern Med. 2014 Mar;174(3):357-68. doi: 10.1001/jamainternmed.2013.13018. PMID 24395196
- [Background] Hofmann SG, Sawyer AT, Witt AA, Oh D. The effect of mindfulness-based therapy on anxiety and depression: A meta-analytic review. J Consult Clin Psychol. 2010 Apr;78(2):169-83. doi: 10.1037/a0018555. PMID 20350028
- [Background] Holzel BK, Lazar SW, Gard T, Schuman-Olivier Z, Vago DR, Ott U. How Does Mindfulness Meditation Work? Proposing Mechanisms of Action From a Conceptual and Neural Perspective. Perspect Psychol Sci. 2011 Nov;6(6):537-59. doi: 10.1177/1745691611419671. PMID 26168376
- [Background] Lorig KR, Sobel DS, Ritter PL, Laurent D, Hobbs M. Effect of a self-management program on patients with chronic disease. Eff Clin Pract. 2001 Nov-Dec;4(6):256-62. PMID 11769298
- [Background] Schuman-Olivier Z, Hoeppner BB, Evins AE, Brewer JA. Finding the right match: mindfulness training may potentiate the therapeutic effect of nonjudgment of inner experience on smoking cessation. Subst Use Misuse. 2014 Apr;49(5):586-94. doi: 10.3109/10826084.2014.850254. PMID 24611853
- [Background] Alegria M, Sribney W, Perez D, Laderman M, Keefe K. The role of patient activation on patient-provider communication and quality of care for US and foreign born Latino patients. J Gen Intern Med. 2009 Nov;24 Suppl 3(Suppl 3):534-41. doi: 10.1007/s11606-009-1074-x. PMID 19842003
- [Background] Neff KD, Germer CK. A pilot study and randomized controlled trial of the mindful self-compassion program. J Clin Psychol. 2013 Jan;69(1):28-44. doi: 10.1002/jclp.21923. Epub 2012 Oct 15. PMID 23070875
- [Background] Wiegner L, Hange D, Bjorkelund C, Ahlborg G Jr. Prevalence of perceived stress and associations to symptoms of exhaustion, depression and anxiety in a working age population seeking primary care--an observational study. BMC Fam Pract. 2015 Mar 19;16:38. doi: 10.1186/s12875-015-0252-7. PMID 25880219
- [Background] Benzo RP. Mindfulness and motivational interviewing: two candidate methods for promoting self-management. Chron Respir Dis. 2013 Aug;10(3):175-82. doi: 10.1177/1479972313497372. PMID 23897933
- [Background] Gawande R, To MN, Pine E, Griswold T, Creedon TB, Brunel A, Lozada A, Loucks EB, Schuman-Olivier Z. Mindfulness Training Enhances Self-Regulation and Facilitates Health Behavior Change for Primary Care Patients: a Randomized Controlled Trial. J Gen Intern Med. 2019 Feb;34(2):293-302. doi: 10.1007/s11606-018-4739-5. Epub 2018 Dec 3. PMID 30511291

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 11 metro-north Boston primary care Patient Centered Medical Homes via print and digital flyers, as well as referrals from primary and mental health care settings confirmed by a primary care provider. 465 participants were recruited.
Pre-assignment Details: All participants received a 60-minute introduction to mindfulness led by an MTPC group leader prior to randomization. The session included a conceptual/experiential mindfulness introduction, inquiry, and digital and print resources. Participants were able to decline study continuation after the 60-minute introduction and before randomization.
Period: Overall Study
Arm/Group | Mindfulness Training for Primary Care | Low-dose Comparator
Started | 92 | 44
Completed | 68 (Completed 8 or 9 week Action Plan Initiation Survey) | 32 (Completed 8 or 9 week Action Plan Initiation Survey)
Not Completed | 24 | 12
Not completed — Lost to Follow-up | 17 | 5
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Partially completed 8 wk or 24 wk survey | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness Training for Primary Care | Low-dose Comparator | Total
Number analyzed (Participants) | 92 | 44 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (12.7) | 40.3 (12.2) | 40.5 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 26 | 89
  Male | 29 | 18 | 47
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic | 17 | 4 | 21
  Ethnicity: Non-Hispanic | 75 | 40 | 115
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 73 | 32 | 105
  Race: Black | 3 | 4 | 7
  Race: Other | 16 | 8 | 24
English as second language [Count of Participants; unit: Participants] | 19 | 5 | 24
Annual Income <$20,000 [Count of Participants; unit: Participants] | 31 | 9 | 40
Marital Status [Count of Participants; unit: Participants]
  Single | 44 | 23 | 67
  Married/cohabitating | 32 | 17 | 49
  Divorced | 13 | 2 | 15
  Widowed | 1 | 1 | 2
  Other | 2 | 1 | 3
Education [Mean (Standard Deviation); unit: years] | 16.6 (3.1) | 15.5 (4.1) | 16.2 (3.4)
Insurance [Count of Participants; unit: Participants]
  Medicaid or Medicare | 12 | 8 | 20
  Subsidized | 39 | 12 | 51
  Private | 39 | 22 | 61
  Other | 2 | 2 | 4
Have practiced meditation before [Count of Participants; unit: Participants] | 56 | 22 | 78
Baseline meditation practice [Mean (Standard Deviation); unit: minutes/day] | 6.8 (10.5) | 4.1 (6.5) | 5.9 (9.4)
DSM-V diagnosis [Count of Participants; unit: Participants]
  Single DSM-V diagnosis | 59 | 30 | 89
  2+ DSM-V diagnosis | 33 | 14 | 47
Primary DSM-V diagnosis [Count of Participants; unit: Participants]
  Major depressive disorder | 27 | 10 | 37
  Generalized anxiety disorder | 16 | 7 | 23
  Anxiety NOS | 14 | 6 | 20
  Adjustment disorder | 11 | 10 | 21
  Other depressive disorder | 9 | 6 | 15
  Other | 15 | 5 | 20
Any PTSD diagnosis [Count of Participants; unit: Participants] | 11 | 1 | 12
Any depression diagnosis [Count of Participants; unit: Participants] | 48 | 19 | 67

OUTCOME MEASURES:

1. Primary Outcome: Action Plan Initiation Survey (APIS-5)
Description: The Action Plan Initiation Survey (APIS-5) is a 5-item self-report questionnaire adapted from a measure used by Guck et al. Participants are asked to indicate how successful they were in meeting a previously set Action Plan by using a 7-point Likert scale from 1 (Not met at all) to 7 (Totally met), with a score of 5 or above indicating successful initiation of the goal. For each unmet goal, patients are asked to further rate the cause of not meeting the goal by using a 7-point Likert rating scale from 1 (Extremely controllable) to 7 (Not at all controllable).
  For this outcome we reported the number of participants in each arm who successfully initiated an Action Plan, as indicated by a score of 5 or above in reporting whether they were able to meet their action plan goal.
Time Frame: Weeks 8-10
Population: Using mixed effects intent-to-treat analysis, we defined non-initiator status as participants who never endorsed greater than 4 or who did not complete the API survey. by week 9. The APIS-5 is analyzed using an intent to treat analysis and missing APIS is considered incomplete action plan initiation.
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness Training for Primary Care | Low-dose Comparator
Number analyzed (Participants) | 92 | 44
Participants | 53 | 14
Statistical Analysis 1: Comparison: Mindfulness Training for Primary Care vs Low-dose Comparator; Test type: Superiority; p = 0.006, Unadjusted bivariate logistic regression; Odds Ratio (OR) = 2.91

2. Primary Outcome: Perceived Stress Scale
Description: The Perceived Stress Scale (PSS) (10 items) measures the degree to which situations in life are stressful. Items are designed to evaluate how overloaded, unpredictable, and uncontrollable one finds one's life. Each item is scored on a 5 point Likert scale from 0 (Never) to 4 (Very often). Scores range from 0-40 with higher scores reflecting worse results (more stress).
Time Frame: Baseline and week 8 (pre to post Intervention)
Population: We conducted a difference-in-differences, ITT, repeated measures analysis using linear mixed effects models
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training for Primary Care | Low-dose Comparator
Number analyzed (Participants) | 92 | 44
score on a scale
  Baseline | 25.0 (6.7) | 24.3 (6.6)
  8 Weeks | 19.9 (6.3) | 20.9 (6.3)
Statistical Analysis 1: Comparison: Mindfulness Training for Primary Care vs Low-dose Comparator; Test type: Superiority; p = 0.19, Mixed Models Analysis; Cohen's d: -0.25

3. Primary Outcome: Patient Reported Outcomes Measurement Information System - Anxiety Short Form (PROMIS-ASF)
Description: The Patient Reported Outcomes Measurement Information System - Anxiety Short Form 8a (PROMIS-ASF) is an 8-item scale used to assess patient-reported health status for anxiety. PROMIS instruments are funded by the National Institutes of Health (NIH) and used to reliably and validly measure patient-reported outcomes for clinical research and practice. Participants are asked to rate their experience of the item in the past seven days on a 5-point Likert scale from 1 (Never) to 5 (Always). The values of the response to each question are summed into a raw score ranging from 8-40. The raw score is then rescaled with use of the PROMIS Assessment Center Scoring Service into a T score, a standardized score with a mean of 50 and a standard deviation (SD) of 10. Higher T-Score reflects worse results (greater symptom severity).
Time Frame: Baseline and week 8 (pre to post Intervention)
Population: We conducted a difference-in-differences, ITT, repeated measures analysis using linear mixed effects models
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training for Primary Care | Low-dose Comparator
Number analyzed (Participants) | 92 | 44
score on a scale
  Baseline | 63.9 (6.9) | 61.9 (6.6)
  8 Weeks | 58.5 (6.6) | 58.9 (6.9)
Statistical Analysis 1: Comparison: Mindfulness Training for Primary Care vs Low-dose Comparator; Test type: Superiority; p = 0.12, Mixed Models Analysis; Cohen's d: -0.36

4. Primary Outcome: Patient Reported Outcomes Measurement Information System - Depression Short Form (PROMIS-DSF)
Description: The Patient Reported Outcomes Measurement Information System - Depression Short Form 8a (PROMIS-DSF) is an 8-item scale used to assess patient-reported health status for depression. PROMIS instruments are funded by the National Institutes of Health (NIH) and used to reliably and validly measure patient-reported outcomes for clinical research and practice. Participants are asked to rate their experience of the item in the past seven days on a 5-point Likert scale from 1 (Never) to 5 (Always). The values of the response to each question are summed into a raw score ranging from 8-40. The raw score is then rescaled with use of the PROMIS Assessment Center Scoring Service into a T score, a standardized score with a mean of 50 and a standard deviation (SD) of 10. Higher T-Score reflects reflect worse results (greater symptom severity).
Time Frame: Baseline and week 8 (pre to post Intervention)
Population: We conducted a difference-in-differences, ITT, repeated measures analysis using linear mixed effects models
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training for Primary Care | Low-dose Comparator
Number analyzed (Participants) | 92 | 44
score on a scale
  Baseline | 59.2 (8.6) | 58.0 (8.6)
  8 Weeks | 53.9 (7.9) | 55.6 (8.0)
Statistical Analysis 1: Comparison: Mindfulness Training for Primary Care vs Low-dose Comparator; Test type: Superiority; p = 0.08, Mixed Models Analysis; Cohen's d: -0.34

5. Secondary Outcome: Five Facet Mindfulness Questionnaire (FFMQ)
Description: The Five Facet Mindfulness Questionnaire (FFMQ) is a 39-item scale that examines five factors that represent aspects of the current empirical conception of mindfulness. These five facets include: "observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience." Participants rate their degree of agreement with each of the items on a Likert-type scale ranging from 1 (Never or very rarely true) to 5 (Very often or always true). Facet scores range from 8-40, with the exception of the nonreactivity facet, which ranges from 7-35. Total scores range from 39-195, with higher scores reflecting higher levels of mindfulness (a better outcome).
Time Frame: Baseline and week 8 (pre to post Intervention)
Population: We conducted a difference-in-differences, ITT, repeated measures analysis using linear mixed effects models
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training for Primary Care | Low-dose Comparator
Number analyzed (Participants) | 92 | 44
score on a scale
  Baseline | 115.8 (18.2) | 115.6 (24.5)
  8 Weeks | 132.0 (16.9) | 119.4 (26.4)
Statistical Analysis 1: Comparison: Mindfulness Training for Primary Care vs Low-dose Comparator; Test type: Superiority; p < 0.001, Mixed Models Analysis; Cohen's d: 0.57

6. Secondary Outcome: Self-Compassion Scale-Short Form (SCS-SF)
Description: The short-form Self-Compassion Scale (SCS-SF) is an abbreviated 12-item form of the original 26-item Self-Compassion Scale. The scale is scored on a 5 point Likert scale (1 = Almost never; 5 = Almost always), and negative subscale items are reverse scored, with higher scores indicating greater levels of self-compassion.
Time Frame: Baseline and week 8 (pre to post Intervention)
Population: We conducted a difference-in-differences, ITT, repeated measures analysis using linear mixed effects models
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training for Primary Care | Low-dose Comparator
Number analyzed (Participants) | 92 | 44
score on a scale
  Baseline | 2.6 (0.67) | 2.6 (0.73)
  8 Weeks | 3.1 (0.65) | 2.8 (0.69)
Statistical Analysis 1: Comparison: Mindfulness Training for Primary Care vs Low-dose Comparator; Test type: Superiority; p = 0.03, Mixed Models Analysis; Cohen's d: 0.41

7. Secondary Outcome: Change in Self-Efficacy for Managing Chronic Disease (SECD-6)
Description: The Self-Efficacy for Managing Chronic Disease Scale (SECD-6) is a 6-item scale that is used to evaluate a participant's ability to self-manage care for a chronic disease. SECD-6 asks participants to rate their confidence in their own ability to do certain activities, on a scale from 1 (not at all confident) to 10 (totally confident). Higher scores indicate better results (higher levels of self-efficacy).
Time Frame: Baseline and week 8 (pre to post Intervention)
Population: We conducted a difference-in-differences, ITT, repeated measures analysis using linear mixed effects models
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training for Primary Care | Low-dose Comparator
Number analyzed (Participants) | 92 | 44
score on a scale
  Baseline | 6.1 (1.9) | 6.2 (2.0)
  8 Weeks | 6.7 (1.6) | 6.5 (1.7)
Statistical Analysis 1: Comparison: Mindfulness Training for Primary Care vs Low-dose Comparator; Test type: Superiority; p = 0.31, Mixed Models Analysis; Cohen's d: 0.15

8. Secondary Outcome: Perceived Control Questionnaire (PCQ)
Description: The Perceived Control Questionnaire (PCQ) is adapted from a 5-item perceived control measure from Jerant et al. and a previously validated survey from Armitage et al. This 5-item scale asks participants to rate their sense of control over chronic illness self-management on a 7-point scale from 1 (None) to 7 (Total). Scores range from 5-35, with higher scores indicating better results (greater sense of control).
Time Frame: Baseline and week 8 (pre to post Intervention)
Population: We conducted a difference-in-differences, ITT, repeated measures analysis using linear mixed effects models
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training for Primary Care | Low-dose Comparator
Number analyzed (Participants) | 92 | 44
score on a scale
  Baseline | 23.5 (4.4) | 23.0 (4.4)
  8 Weeks | 25.3 (4.2) | 23.8 (4.3)
Statistical Analysis 1: Comparison: Mindfulness Training for Primary Care vs Low-dose Comparator; Test type: Superiority; p = 0.26, Mixed Models Analysis; Cohen's d: 0.22

9. Secondary Outcome: Difficulty in Emotion Regulation Scale (DERS)
Description: The Difficulties in Emotion Regulation (DERS) Scale is a 36-item self-report scale designed to assess emotional dysregulation. Participants are asked to rate how often they have emotional dysregulation on a 5-point Likert scale from 1 (almost never [0-10%]) to 5 (almost always [91-100%]). The scale assess 6 aspects of emotional dysregulation: non-acceptance of emotional responses, difficulties engaging in goal directed behavior, impulse control difficulties, lack of emotional awareness (reverse-scored), limited access to emotion regulation strategies, and lack of emotional clarity. Total scores range from 5-180, with higher scores indicating worse results (more difficulty in emotional regulation).
Time Frame: Baseline and week 8 (pre to post Intervention)
Population: We conducted a difference-in-differences, ITT, repeated measures analysis using linear mixed effects models
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training for Primary Care | Low-dose Comparator
Number analyzed (Participants) | 92 | 44
score on a scale
  Baseline | 76.1 (23.0) | 72.2 (23.2)
  8 Weeks | 60.2 (21.8) | 68.8 (21.8)
Statistical Analysis 1: Comparison: Mindfulness Training for Primary Care vs Low-dose Comparator; Test type: Superiority; p < 0.001, Mixed Models Analysis; Cohen's d: -0.58

10. Secondary Outcome: Multidimensional Assessment of Interoceptive Awareness (MAIA)
Description: The Multidimensional Assessment of Interoceptive Awareness (MAIA) is a 32-item self-report scale designed to assess 8 aspects of interoceptive awareness : noticing, not-distracting, not-worrying, attention regulation, emotional awareness, self-regulation, body listening, and trusting. Participants are asked to rate their awareness of interoceptive experiences on a 6-point Likert scale from 0 (Never) to 5 (Always). Each subscale has 3-7 items, and scores are obtained by reverse coding items 5, 6, 7, 8, 9, and then taking the average of items in each scale. Scores range from 0-5, with higher scores indicating better results (greater interoception).
Time Frame: Baseline and week 8 (pre to post Intervention)
Population: We conducted a difference-in-differences, ITT, repeated measures analysis using linear mixed effects models
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training for Primary Care | Low-dose Comparator
Number analyzed (Participants) | 92 | 44
score on a scale
  Baseline | 2.4 (0.73) | 2.5 (0.73)
  8 Weeks | 3.1 (0.64) | 2.6 (0.69)
Statistical Analysis 1: Comparison: Mindfulness Training for Primary Care vs Low-dose Comparator; Test type: Superiority; p < 0.001, Mixed Models Analysis; Cohen's d: 0.75

ADVERSE EVENTS:
Time Frame: Participants completed a self-reported adverse events form during weeks 8 and 24. Adverse events were further collected during engagement phone calls during weeks 2, 4 6, and 8 using a combination of checklist and open-ended questions.
Description: An adverse event is any untoward medical occurrence in a subject during participation in the clinical study. An adverse finding can include a sign, symptom, abnormal assessment (from vital signs or brain imaging), or any combination of these. AEs will be labeled according to severity based on their impact on the patient on the patient's well-being: "mild" if it does not have major impact, "moderate" if it causes some minor inconvenience, and "severe" if it causes substantial disruption.
Arm/Group | Mindfulness Training for Primary Care | Low-dose Comparator
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/44
Serious Adverse Events (participants affected / at risk) | 4/92 | 0/44
Other Adverse Events (participants affected / at risk) | 8/92 | 4/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mindfulness Training for Primary Care (N=92) | Low-dose Comparator (N=44)
Diagnosed with colon cancer (Gastrointestinal disorders) | 1 (1) | NA
Psychiatric hospitalization, hypomanic episode (Psychiatric disorders) | 1 (1) | NA — Worsening of underlying condition
Psychiatric hospitalization, increased PTSD symptoms (Psychiatric disorders) | 1 (1) | NA — Worsening of underlying condition
Psychiatric hospitalization, suicidal ideation (Psychiatric disorders) | 1 (1) | NA — Worsening of underlying condition
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mindfulness Training for Primary Care (N=92) | Low-dose Comparator (N=44)
Back injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
ED visit for alcohol abuse (Psychiatric disorders) | 1 (2) | 0 (0)
Binge drinking (Psychiatric disorders) | 0 (0) | 1 (1)
Motor vehicle accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Motor vehicle accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ED visit after alleged sexual assault (Social circumstances) | 1 (1) | 0 (0)
Flashback during MTPC All-Day Session (Psychiatric disorders) | 1 (1) | 0 (0) — Participant calmed himself, finished the session, and received consultation from group leaders
Increased Anxiety during Open Awareness Practice (Psychiatric disorders) | 1 (1) | 0 (0) — Participant consulted with the group leader and continued participating
ED visit due to hearing loss, ear pain, tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Corneal abrasion (Eye disorders) | 1 (1) | 0 (0)
Admission for flu and UTI (Renal and urinary disorders) | 0 (0) | 1 (1) — This event was reported to CHA IRB, which responded on 5/17/2018 that this event is not considered an SAE

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/00/NCT03265600/Prot_SAP_000.pdf